CLINICAL TRIAL: NCT03304769
Title: Virtual Reality Distraction During Pediatric Intravenous Line Placement: A Prospective Randomized Comparison Study
Brief Title: Virtual Reality Distraction During Pediatric Intravenous Line Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Collaborators: Seton Healthcare Family (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ASalinas
Record Dates: First submitted 2017-09-28; First posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Pediatric IV Placement; Virtual Reality Distraction
Keywords: Virtual Reality Distraction; Pediatric IV placement

STUDY DESIGN:
Intervention Model Description: Selected from a single-site level one pediatric emergency department. Pediatric patients aged 4-17 years requiring an IV. Random number generator used to decide which patients will be using VR and which will have standard IV placement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV placement no Virtual reality (No Intervention): Patient will have IV placed in traditional manner, with no virtual reality headset
- IV placement with Virtual Reality (Experimental): Patient will have IV placed with Virtual Reality headset distraction
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Virtual Reality Headset applied to the patient during placement of IV. Control is patient group without headset applied.
  Arms: IV placement with Virtual Reality

SUMMARY:
This study aims to prospectively investigate the use of virtual reality headsets on the placement of IVs in a pediatric emergency department, by comparing the first stick success rate, total number of attempts, and the time to successful IV placement between patients who use virtual reality headset technology during the placement and those who receive the standard of care IV placement when child life ( individuals with special training in aiding and augmenting pediatric coping skills) is not available. The investigators will also compare the patient and parent perception of pain and anxiety associated with the IV placement in both study groups. Finally, by detailing which medications have been given prior to use of the VR for IV placement the investigators may evaluate for possible synergistic effects of VR with prior medication administration.

DETAILED DESCRIPTION:
Children often describe procedures involving needles as the most stressful portion of the hospital experience. 1,2 Many studies involving the perception of pain have highlighted the importance of attention for the perception of pain, and, conversely, the benefit of distraction for decreasing pain perception. 3,4 Virtual reality technologies (VR) have been shown to mitigate the experience of pain and anxiety in patients undergoing procedures in a number of different ways. 5,6 While small studies have demonstrated the use of VR to be effective in diminishing pain during intravenous (IV) placement for outpatient imaging in pediatric patients aged 8-12, there have not been large-scale studies assessing the use of VR during IV placement in the Pediatric Emergency Department. 7 Studies examining the use of VR during venipuncture and IV placement also frequently focus on self-reported or parent-reported pain, rather than objectively quantifying number of IV sticks and time to successful IV placement.8 Additionally, the pediatric age ranges which benefit from VR have not been well-established, with some studies citing benefits only in patients over 10 years of age, and others showing improvements in all age groups.7,9,10

This study aims to prospectively investigate the use of virtual reality headsets on the placement of IVs in a pediatric emergency department, by comparing the first stick success rate, total number of attempts, and the time to successful IV placement between patients who use virtual reality headset technology during the placement and those who receive the standard of care IV placement when child life ( individuals with special training in aiding and augmenting pediatric coping skills) is not available. The investigators will also compare the patient and parent perception of pain and anxiety associated with the IV placement in both study groups. Finally, by detailing which medications have been given prior to use of the VR for IV placement the investigators may evaluate for possible synergistic effects of VR with prior medication administration.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 4-17 years
* Requiring IV placement
* Child Life unavailable

Exclusion Criteria:

* Previous enrollment in the study
* Physically/ developmentally unable to tolerate headset
* Skin/eye pathology
* Critically ill patient
* Language other than English or Spanish
* Student Nurse placing IV

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 116 (Estimated)
Dates: Start 2017-09-28 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Successful IV placement with first attempt | 6 months
  success in first attempt in VR group vs non VR group

SECONDARY OUTCOMES:
number of attempts before successfully establishing IV | 6 months
  number of attempts before successful IV placement in VR group vs non VR group
time to establishing successful IV | 6 months
  time to establishing successful IV in VR group vs non VR group
Pre vs Post FACES revised pain scale parents | 6 months
  Pre vs Post FACES pain scale in VR group vs non VR group
Pre vs Post FACES revised pain Scale patients | 6 months
  Pre vs Post FACES pain scale in VR group vs non VR group
Pre vs Post Likert-Type Anxiety Scale - parents | 6 months
  Pre vs Post Likert-Type Anxiety Scale of parents in VR group vs non VR group
Pre vs Post Likert-Type Anxiety Scale- patients | 6 months
  Pre vs Post Likert-Type Anxiety Scale of patients in VR group vs non VR group
age range of patients that tolerate VR | 6 months
  Which of evaluated age range of 4-17 years tolerate VR placement

CONTACTS AND LOCATIONS:
Locations (1):
- Dell Children's Medical Center of Central Texas, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No